CLINICAL TRIAL: NCT04294264
Title: TAS-102 in Combination With Oxaliplatin (TAS-OX) for Refractory Metastatic Colorectal Cancer
Brief Title: TAS-102 and Oxaliplatin for the Treatment of Refractory Stage IV Colon Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Howard S. Hochster, MD, Associate Director for Clinical Research Medical Oncology, Rutgers Cancer Institute of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro2018001469; NCI-2020-00871 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Pro2018001469; 071801 (Other: Rutgers Cancer Institute of New Jersey); P30CA072720 (NIH)
Record Dates: First submitted 2020-03-02; First posted 2020-03-04 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Metastatic Colorectal Carcinoma; Recurrent Colon Carcinoma; Refractory Colorectal Carcinoma; Stage IV Colon Cancer AJCC v7; Stage IVA Colon Cancer AJCC v7; Stage IVB Colon Cancer AJCC v7
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — Oxaliplatin; Trifluridine; trifluridine tipiracil drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (TAS-102, oxaliplatin) (Experimental): Patients receive TAS-102 PO BID on days 1-5 and oxaliplatin IV over 2 hours on day 1. Cycles repeat every 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Oxaliplatin; Drug: Trifluridine and Tipiracil Hydrochloride

INTERVENTIONS:
Drug: Oxaliplatin — Given IV
  Other Names: 1-OHP; Ai Heng; Aiheng; Dacotin; Dacplat; Diaminocyclohexane Oxalatoplatinum; Eloxatin; Eloxatine; JM-83; Oxalatoplatin; Oxalatoplatinum; RP 54780; RP-54780; SR-96669
Drug: Trifluridine and Tipiracil Hydrochloride — Given PO
  Other Names: Lonsurf; TAS 102; TAS-102; Tipiracil Hydrochloride Mixture with Trifluridine; Trifluridine/Tipiracil; Trifluridine/Tipiracil Hydrochloride Combination Agent TAS-102

SUMMARY:
This phase II trial studies how well TAS-102 and oxaliplatin work in treating patients with stage IV colon cancer. Drugs used in chemotherapy, such as TAS-102 and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Overall response rate (ORR).

SECONDARY OBJECTIVES:

I. Progression free survival (PFS). II. Overall survival (OS). III. Disease control rate (DCR). IV. Duration of response. V. Safety and tolerability.

OUTLINE:

Patients receive trifluridine and tipiracil hydrochloride (TAS-102) orally (PO) twice daily (BID) on days 1-5 and oxaliplatin intravenously (IV) over 2 hours on day 1. Cycles repeat every 14 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed stage IV colon cancer (American Joint Committee on Cancer [AJCC] 7th edition) that has progressed after standard therapy that included fluorouracil (5-FU), irinotecan, oxaliplatin, bevacizumab (unless contraindicated) and an anti-EGFR antibody, if RAS wild type. Patients who could not tolerate standard agents because of unacceptable, but reversible toxicity necessitating their discontinuation will be allowed to participate
* Patients who had received adjuvant chemotherapy and had recurrence during or within 6 months of completion of the adjuvant chemotherapy will be allowed to count the adjuvant therapy as one chemotherapy regimen
* Progression of disease must be documented on the most recent scan
* Presence of measurable disease
* RAS mutation and mismatch repair deficiency (MMR) status must be determined (or tissue availability for testing if not already determined)
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Life expectancy of at least 3 months
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L
* Hemoglobin >= 9 g/dL
* Platelets (PLT) >= 75 x 10^9/L
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 5 x upper limit of normal (ULN)
* Adequate contraception if applicable
* Women who are nursing and discontinue nursing prior to enrollment in the program
* Ability to take oral medication (i.e., no feeding tube)
* Patient able and willing to comply with study procedures as per protocol
* Patient able to understand and willing to sign and date the written voluntary informed consent form (ICF) at screening visit prior to any protocol-specific procedures

Exclusion Criteria:

* Patients who have previously received TAS-102
* Grade 2 or higher peripheral neuropathy (functional impairment)
* Symptomatic central nervous system (CNS) metastases requiring treatment
* Other active malignancy within the last 3 years (except for non-melanoma skin cancer or a non-invasive/in situ cancer)
* Pregnancy or breast feeding
* Current therapy with other investigational agents
* Active infection with body temperature >= 38 degree Celsius (C) due to infection
* Major surgery within prior 4 weeks (the surgical incision should be fully healed prior to drug administration)
* Any anticancer therapy within prior 3 weeks of first dose of study drug
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to TAS-102
* Current therapy with other investigational agents or participation in another clinical study or any investigational agent received within prior 4 weeks
* Grade 3 or higher hypersensitivity reaction to oxaliplatin, or grade 1-2 hypersensitivity reaction to oxaliplatin not controlled with pre-medication
* Has unresolved toxicity of greater than or equal to Common Terminology Criteria for Adverse (CTCAE) grade 2 attributed to any prior therapies (excluding anemia, alopecia, skin pigmentation, and platinum-induced neurotoxicity)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-02-12 (Actual); Primary Completion 2024-03-27 (Actual); Study Completion 2026-03-27 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | Up to 2 years
  Response rate is defined as the percentage of subjects with a confirmed complete response (CR) or partial response (PR) by investigator assessment as per Response Evaluation Criteria in Solid Tumors (RECIST) criteria, version 1.1. Response rate will be calculated by dose level. Descriptive statistics will be used to analyze efficacy data using historical data as reference.

SECONDARY OUTCOMES:
Progression free survival | From the date of start of treatment to the date of first documented progression or any cause of death during the study, assessed up to 2 years
  Progression will be assessed by a computed tomography CT scan according to RECIST criteria version 1.1. This criterion will be estimated by the Kaplan-Meier method. Patients who have not progressed or died at the time of analysis will be censored at the time of their latest follow-up with clinically stable disease.
Overall survival | Up to 2 years
Disease control rate | Up to 2 years
Duration of response | Up to 2 years
  Response rate will be calculated by dose level. Descriptive statistics will be used to analyze efficacy data using historical data as reference.
Incidence of adverse events | Up to 28 days post treatment
  All recorded adverse events will be listed and tabulated by system organ class and dose level. Will utilize the Cancer Therapy Evaluation Program Common Toxicity Criteria (CTC) version 5.0 for toxicity and adverse event reporting.

CONTACTS AND LOCATIONS:
Overall Officials: Howard S Hochster, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (6):
- United States (6):
  - Trinitas Hospital and Comprehensive Cancer Center, Elizabeth, New Jersey
  - RWJBarnabas Health - Monmouth Medical Center Southern Campus, Lakewood, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - RWJBarnabas Health - Monmouth Medical Center, Long Branch, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - RWJBarnabas Health - Community Medical Center, Toms River, New Jersey

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-09-13): https://cdn.clinicaltrials.gov/large-docs/64/NCT04294264/ICF_000.pdf